CLINICAL TRIAL: NCT05098821
Title: Pattern Recognition of Immune Cells in Atopic Dermatitis Patients Receiving Dupilumab
Brief Title: Extrinsic and Intrinsic Factors in Atopic Dermatitis Upon Systemic Immune Modulation
Acronym: AD-Sys
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Sanofi (Industry); LEO Pharma (Industry)
Responsible Party: Principal Investigator, Margitta Worm, Prof. Dr. med. Margitta Worm, Charite University, Berlin, Germany
Other Study IDs: PRI-ADD
Record Dates: First submitted 2021-10-20; First posted 2021-10-28 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Atopic Dermatitis
Keywords: dupilumab; pattern recognition; immune cells
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dupilumab treated Patients: Patients with atopic dermatitis with indication for dupilumab treatments will be observed
  Interventions: Other: not applicable, observational study

INTERVENTIONS:
Other: not applicable, observational study — Patients undergoing systemic therapy according to international accepted guidelines for the therapy of atopic dermatitis, observational study

SUMMARY:
Currently, patients with moderate to severe atopic dermatitis are treated with dupilumab if unresponsive to topical treatment. However, not all patients who suffer from atopic dermatitis respond similarly to this treatment. Pattern recognition of immune cells (PRI) is an efficient method to screen patients to allow a more personalized therapy.

The main aim of this scientific explorative study is to unravel the changes in peripheral blood immune cell compositions in patients with atopic eczema undergoing dupilumab treatment. This allows the identification of phenotypes of treatment responders and non-responders and possible approaches of treatment modifications for non-responders.

DETAILED DESCRIPTION:
A better understanding of the pathology of atopic dermatitis could lead to the development of new therapeutic strategies for this disease and contribute to better and more targeted disease management - an advantage for all patients with atopic dermatitis.

The PRI is a new bioinformatic analysis strategy that allows in-depth data analysis from flow cytometry with multiple variables. This facilitates the identification of meaningful T cell subpopulations, which are differentially abundant between two groups to predict responders and non-responders prior to dupilumab treatment.

Peripheral blood will be collected before, 4 weeks, 8 weeks, and 16 weeks after initiating the systemic treatment with dupilumab to identify recognition patterns/markers on the T cells. Therefore, a predefined multicolor flow cytometry panel was developed to analyse lineage, differentiation and activation markers.

Patients will receive a systemic therapy (dupilumab 600 mg loading dose, followed by 300 mg in two weeks intervals). Follow up visits will be performed every 3 months starting from the second visit (2nd visit will take place 4 weeks after initiating Dupilumab treatment).

The blood samples that are taken as part of this scientific study are pseudonymized in the research laboratories and stored for a period of 5 years after the end of this study or the publication of the results and destroyed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Diagnosis of atopic dermatitis for ≥1 year
* Inadequate response to treatment with topical medications
* Confirmed dupilumab treatment

Exclusion Criteria:

* Age below 18
* Known or suspected allergy or reaction to any component of the dupilumab formulation
* Known active allergic or irritant contact dermatitis that is likely to interfere with the assessment of the severity of AD
* Severe conjunctivitis or blepharitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with moderate to severe atopic dermatitis presenting in the clinic of Dermatology, Charité - Universitätsmedizin Berlin, Germany
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of T-cell inflammatory markers | 1 year
  Identification of at least one pattern recognition profile showing a strong association with responder status to dupilumab therapy

SECONDARY OUTCOMES:
Different T-cell pattern with dupilumab therapy | 1.5 years
  Time in which the pattern of T-cell modulation after initiation of dupilumab therapy (measured using PRI) shows significant differences from the baseline.
Assign recognition patterns to clinical symptoms | 3 months
  Association of recognition patterns with clinical symptoms of atopic dermatitis (measured using Cramer's V > 0.5) with a specific interest in conjunctivitis, pruritus, asthma and herpes infections.
Connection of molecular profile and phenotype | 3 months
  Classification and clustering of at least two molecular profiles of peripheral blood immune cells in relation to phenotypes of atopic dermatitis (Cramer's V either with association to IgE levels or early/late onset AD).

CONTACTS AND LOCATIONS:
Locations (1):
- Dpt of Dermatology and Allergology, Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided